CLINICAL TRIAL: NCT07371065
Title: A Randomized, Double-blind, Dose-escalation Phase I Clinical Study to Evaluate the Safety, Tolerability, be Consistency and Food Effects of LY03021 Tablets in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Food Effects of LY03021 in Healthy Chinese Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03021/CT-CHN-101
Record Dates: First submitted 2025-12-05; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03021 group (Experimental): Orally only once
  Interventions: Drug: LY03021
- Placebo (Sham Comparator): Orally only once
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LY03021 — Orally only once
  Arms: LY03021 group
Drug: placebo — Orally only once
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized withdrawal, double-blind, parallel, placebo-controlled design clinical trial of Toludesvenlafaxine Hydrochloride Extended-Release Tablets to evaluate the long-term efficacy and safety in the treatment of Chinese patients with depression.

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily participate in and sign the informed consent form after understanding the purpose, content, process and possible risks of the trial;
2. Healthy male/female volunteers between 18 and 45 years of age, inclusive, at the time of signing the informed consent form;
3. Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) 18.5 kg/m2~ 28.0 kg/m2 (including the boundary value) at screening;
4. Be able to communicate well with the Investigator and comply with the lifestyle restrictions specified in the protocol and various requirements of the clinical trial (scheduled visits, laboratory tests and other trial procedures).

Exclusion Criteria:

1. Known to have a history of allergy to any component of the Investigational product or similar drugs, or allergic constitution (previous allergy to two or more foods or drugs);
2. The subject has a current or past medical history that may affect the clinical trial or dysfunction, including but not limited to a past or present respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry, dermatology and any other clinically significant disease or chronic disease; or any other disease that may interfere with the test results;
3. Any surgical conditions or conditions that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a risk to the subjects participating in the trial, including a history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding, etc.;
4. Subjects with current or past mental disorders and brain dysfunction, or at risk of suicide according to Columbia-Suicide Severity Rating Scale (C-SSRS), or having a suicide risk at the discretion of the Investigator, , or with a history of self-mutilation;
5. History of substance abuse or positive result in urine drug screening within 1 year prior to dosing;
6. History of alcohol abuse (defined as more than 14 standard units of alcohol per week, 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine) or positive breath test results within 1 year before dosing;
7. Subjects who have a history of surgery within 3 months before dose administration, or have not recovered from surgery, or have an anticipated surgical planning during the trial;
8. Those who have participated in other clinical trials within 3 months before dose administration (including drug and medical device clinical trials, the time is based upon the last visit);
9. Blood donation or blood loss ≥ 400 mL within 3 months before dose administration, or blood donation or blood loss ≥ 200 mL within one month, or having a history of using blood products;
10. Pregnant and lactating women; and those who refuse to take effective contraception measures (such as abstinence, intrauterine device or condom with intravaginal spermicide, etc.) during the study period and within 28 days after the end of the study, or have the plan to donate sperm or eggs;
11. Abnormalities in vital signs, laboratory tests and 12-lead electrocardiogram (ECG) , and clinically significant as judged by the Investigator, for example:

    QTc > 450 ms for males and > 460 ms for females, Friericia's correction; Resting pulse rate < 55 beats/min or > 100 beats/min; systolic blood pressure < 90 mmHg or ≥ 140 mmHg; diastolic blood pressure < 60 mmHg or ≥ 90 mmHg;
12. Use of the following medications or treatments prior to dosing:

    Use of any prescription medication within 28 days prior to dosing; Use of any over-the-counter medications, including health products, within 7 days prior to dosing;
13. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), syphilis serum reaction (Trust) non-negative;
14. The average daily smoking of ≥ 5 cigarettes within 3 months before dose administration;
15. Those who have special requirements for food and cannot abide by the unified diet or have dysphagia;
16. Consumption of food or beverages containing grapefruit and/or pomelo within 7 days prior to dosing;
17. Consumption of xanthine-rich foods or beverages (such as tea, coffee, cola or chocolate) within 3 days before dose administration;
18. Poor compliance or any condition that is considered as unsuitable for the study participation by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Day 12

SECONDARY OUTCOMES:
PK parameters: Cmax | Day 12
PK parameters: Tmax | Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- No. 604 Lingling Road, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No